CLINICAL TRIAL: NCT01965756
Title: A Phase II Trial to Study the Effect of Metformin on AD Biomarkers: A Randomized Placebo Controlled Crossover Pilot Study of Metformin Effects on Cognitive, Physiological and Biochemical Biomarkers of MCI and Dementia Due to AD
Brief Title: Effect of Insulin Sensitizer Metformin on AD Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPenn-AHAF_A2012116
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer's Disease; Vascular Dementia; Dementia; Memory Impairment
Keywords: Alzheimer's Disease; Vascular Dementia; Dementia; Memory Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Dementia; Memory Disorders | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This pilot study used a randomized, double-blinded, placebo-controlled 16 week crossover design to examine the effects of metformin on biochemical, neurophysiological, and cognitive biomarkers of AD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin, Then Placebo (Experimental): Participants first received metformin for 8 weeks, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached. After 8 weeks, subjects were switched to matching placebo for an additional 8 weeks.
  Interventions: Drug: Metformin; Drug: Placebos
- Placebo, Then Metformin (Experimental): Participants first received placebo for 8 weeks. After 8 weeks, subjects were switched to metformin, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached.
  Interventions: Drug: Metformin; Drug: Placebos

INTERVENTIONS:
Drug: Metformin
Drug: Placebos

SUMMARY:
Alzheimer's disease (AD) is a neurodegenerative disorder characterized by progressive loss of memory and other cognitive functions. It is the most common cause of dementia in older adults, affecting approximately 18 million people worldwide, including almost 500,000 in the Philadelphia tri-state area. After age 65, the incidence of AD rises exponentially, doubling every five years. By age 85, almost half of us will have AD. In 2030, as many as 7.7 million Americans could have AD, and by 2050 this number could rise to 11-16 million people. The annual cost of AD in the United States is about $200 billion. AD-related medical complications are among the most common causes of death in the elderly population. Despite these alarming statistics, a "cure" for AD may not be essential since delaying the onset of AD by just 5 years could have a profound impact on this disorder by reducing the incidence and cost of AD by 50% between now and 2050.

AD is difficult to recognize in its earliest stages, in which the principal complaint is typically an increase in episodes of forgetfulness. This stage is now commonly referred to as mild cognitive impairment (MCI). Neuroimaging and CSF biomarkers have demonstrated good accuracy in predicting which MCI patients later "convert" to AD and which tend to remain stable or revert to more normal cognition. The diagnosis of AD itself is made when increased loss of memory and other cognitive abilities (eg, language, praxis, and executive function) affect daily functioning. As the symptoms of dementia inevitably worsen, patients may become incapable of even basic activities such as feeding and dressing themselves. The disease course often spans more than a decade, creating a vast social and financial burden on society and extracting an immeasurable emotional toll on family members.

Clinical and preclinical evidence is accumulating that brain insulin resistance may play a role in the pathogenesis and/or progression of Alzheimer's disease and that ameliorating insulin action in the brain may benefit cognition symptomatically and modify disease pathology.

ELIGIBILITY:
Inclusion Criteria:

* • Ages 55-80.

  * 2 Sex distribution: male and female
  * Diagnosis of MCI due to AD127 or early dementia due to AD128 with: a) age 55 - 80, b) complaint of cognitive decline, c) abnormal performance on the Logical Memory subtest of the Wechsler Memory Scale, d) MMSE > 21, e) CDR 0.5-1, f) positive topographic (MRI, FDG-PET) or molecular (CSF, amyloid imaging) biomarker consistent with AD, and g) no history of diabetes or other exclusions.
  * Fluent in English or Spanish
  * Education >5, literate, and/or good working history that precludes consideration of mental retardation
  * Visual and auditory acuity sufficient for neuropsychological testing and auditory evoked potential EEG
  * Geriatric Depression Scale < 6
  * Modified Hachinski Ischemic Score < 4
  * No major health issues or diseases expected to interfere with the study
  * Willing to complete all baseline assessments and study procedures
  * Stable on all permitted medications for 8 weeks
  * Not pregnant, lactating or of child-bearing potential (women must be >2 years post-menopausal or surgically sterile)
  * No history of diabetes
  * Fasting blood glucose <126 and/or HgbA1c < 6.4
  * Study partner with frequent contact with patient willing to accompany patient to visits and complete partner study forms
  * No contraindication to metformin

Exclusion Criteria:

* • Any CNS disease other than suspected incipient AD, such as clinical stroke, brain tumor, normal pressure hydrocephalus, brain tumor, multiple sclerosis, significant head trauma with persistent neurological of cognitive deficits or complaints, Parkinson's disease, frontotemporal dementia, or other neurodegenerative diseases

  * Screening/baseline MRI scans with evidence of infarction or other focal lesions in critical memory structures that may be related to cognitive dysfunction
  * Major active psychiatric illness (e.g., depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) within the previous year
  * History of alcohol or other substance abuse or dependence within the past two years
  * Pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body or claustrophobia that would preclude MRI scanning
  * History of past or current diabetes, pancreatic or liver disease, renal disease
  * Any significant systemic illness or unstable medical condition that could affect compliance with study
  * Laboratory abnormalities in B12, TFTs, RPR, Lyme or other common lab parameters that might contribute to cognition or participation in study
  * Coagulopathy or anti-coagulant therapy (such as coumadin) increasing the risk for LP resulting in PT/PTT and INR within 1.5 standard deviations over the upper normal limit.
  * Compromised renal function at screening as determined by creatinine clearance <30mL/min based on Cockcroft-Gault calculation
  * Liver dysfunction at screening as evidenced by alanine transaminase (ALT/SGPT) values > 2X upper limit of normal or aspartate transaminase (AST/SGOT) values > 3X or total bilirubin > 2X.
  * Has received acetylcholinesterase inhibitor and/or memantine and/or any other medicine that affects the central nervous system for less than 4 months or has less than 2 months stable therapy on these treatments by baseline visit.
  * Current use of specified medications with psychoactive properties that deleteriously affect cognition (e.g., certain antidepressants, anticholinergics, anti-histamines, antipsychotics, sedative hypnotics, anxiolytics)
  * Use of investigational agents one month prior to entry and for the duration of the trial
  * Exceptions to these guidelines may be considered on a case-by-case basis at the discretion of the protocol director.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12-22 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Arnold, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Penn Memory Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Weinberg MS, He Y, Kivisakk P, Arnold SE, Das S. Effect of Metformin on Plasma and Cerebrospinal Fluid Biomarkers in Non-Diabetic Older Adults with Mild Cognitive Impairment Related to Alzheimer's Disease. J Alzheimers Dis. 2024;99(s2):S355-S365. doi: 10.3233/JAD-230899. PMID 38160357
- See also: Penn Memory Center — http://www.pennadc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin, Then Placebo (Treatment Sequence A, 0 to 16 Weeks): Participants first received metformin for 8 weeks, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached. After 8 weeks, subjects were switched to matching placebo for an additional 8 weeks.
- Placebo, Then Metformin (Treatment Sequence B, 0 to 16 Weeks): Participants first received placebo for 8 weeks. After 8 weeks, subjects were switched to metformin, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached.
Period: Overall Study
Arm/Group | Metformin, Then Placebo (Treatment Sequence A, 0 to 16 Weeks) | Placebo, Then Metformin (Treatment Sequence B, 0 to 16 Weeks)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (7.40) | 71.1 (6.57) | 70.1 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
HbA1c [Mean (Standard Deviation); unit: percentage] | 5.5 (0.221) | 5.37 (0.236) | 5.44 (0.232)
Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 90.5 (8.77) | 90.9 (14.1) | 90.7 (11.4)
Clinical Dementia Rating - Global (Composite) Score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Dementia Rating (CDR) is a numeric scale used to quantify the severity of symptoms of dementia. A qualified health professional assesses a patient's cognitive and functional performance in six areas: memory, orientation, judgment & problem solving, community affairs, home & hobbies, and personal care. Scores in each of these are combined to obtain a composite score ranging from 0 through 3, with 3 being most severe/impaired. Possible composite rating scores include 0, 0.5, 1, 2, and 3.
  units on a scale | 0.5 (0) | 0.8 (0.789) | 0.658 (.579)

OUTCOME MEASURES:

1. Primary Outcome: Word List Memory Total - ADAS-cog
Description: Alzheimer's Disease Assessment Scale- Cognitive Sub scale (ADAS-COG). Three trials of 10 words each (30 words total)
Time Frame: 16 weeks (total) - measured at baseline, week 8 (crossover), and week 16
Measure: Mean (Standard Deviation); unit: Words recalled
Groups:
- Placebo, Then Metformin: Participants first received placebo for 8 weeks. After 8 weeks, subjects were switched to metformin for 8 weeks, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached.
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin
Number analyzed (Participants) | 10 | 10
Words recalled
  Baseline | 14.35 (3.96) | 14.7 (3.33)
  Week 8 | 15.1 (4.48) | 14.67 (3.74)
  Week 16 | 14.71 (5.29) | 15.5 (5.72)

2. Secondary Outcome: Trails-B
Description: Standard Trails-B assessment, in which subject is asked to begin at Number 1 and draw a line to Letter A, then to Number 2, then to Letter B, then so forth until he/she reaches the END, without lifting their pencil. They should draw the line as fast as possible, and are timed (in seconds).
Time Frame: 16 weeks- measured at baseline, week 8 (crossover), and week 16
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Metformin, Then Placebo: Participants first received metformin for 8 weeks, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached. After 8 weeks, subjects were switched to matching placebo for an additional 8 weeks.
  Participants first received placebo for 8 weeks. After 8 weeks, subjects were switched to metformin, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached.
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin
Number analyzed (Participants) | 10 | 10
Seconds
  Baseline | 164.28 (101.22) | 186.7 (83.42)
  Week 8 | 164 (95.72) | 170.86 (88.2)
  Week 16 | 170.5 (99.99) | 161.8 (91.3)

3. Other Pre Specified Outcome: Cerebrospinal Fluid Amyloid Beta Concentration
Time Frame: baseline and 8 weeks
Population: CSF was only collected from all participants at baseline and again at week 8 (total of two lumbar punctures). This was pre-specified in the protocol, to ensure adequate tolerability for subjects (total of two lumbar punctures, rather than three). Thus, there is a maximum of 10 data points for each category: 10 for MET-->PBO, and 10 for PBO-->MET
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin
Number analyzed (Participants) | 10 | 10
pg/mL
  Baseline | 254.90 (90.38) | 409.01 (145.46)
  Week 8 | 266.73 (26.70) | 424.45 (117.39)

4. Other Pre Specified Outcome: Cerebrospinal Fluid Total Tau Concentration
Time Frame: baseline and 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Metformin, Then Placebo: Participants first received metformin for 8 weeks, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached. After 8 weeks, subjects were switched to matching placebo for an additional 8 weeks.
  Metformin
  Placebos
- Placebo, Then Metformin: Participants first received placebo for 8 weeks. After 8 weeks, subjects were switched to metformin, according to the following dosing schedule: 500 mg by mouth daily for 1 week, then daily dose (in divided doses) increased by 500 mg per week until a maximum of 2000 mg/d (1000mg twice daily) was reached.
  Metformin
  Placebos
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin
Number analyzed (Participants) | 10 | 10
pg/mL
  Baseline | 554.05 (217.29) | 556.14 (361.57)
  Week 8 | 588.53 (180.02) | 554.47 (356.44)

5. Other Pre Specified Outcome: Cerebrospinal Fluid Phosphorylated Tau Concentration
Time Frame: baseline and 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin
Number analyzed (Participants) | 10 | 10
pg/mL
  Baseline | 63.44 (26.95) | 64.62 (23.94)
  Week 8 | 68.12 (15.56) | 64.10 (26.17)

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Groups:
- Metformin: This group includes subjects treated with metformin for the first 8 weeks of the study, as well as subjects treated with metformin during the second 8 weeks of the study.
- Placebo: This group includes subjects treated with placebo for the first 8 weeks of the study, as well as subjects treated with placebo during the second 8 weeks of the study.
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=20) | Placebo (N=20)
Elevated plasma lactate level (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Treatment with metformin has been associated with increased risk for lactic acidosis. As such, serum lactate levels were collected throughout the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No